CLINICAL TRIAL: NCT01786122
Title: PHYSICAL EXERCISE TO IMPROVE THE QUALITY OF LIFE OF CANCER PATIENTS DURING TREATMENT PROCESS: EFICANCER STUDY
Brief Title: Clinical Trial: Effectiveness and Efficiency of Physical Exercise in Cancer Patients
Acronym: EFICANCER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Gonzalo Grandes, Family Medicine specialist, master in epidemiology; Head of the Research Unit of Family Medicine of Bizkaia, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EFICANCER PI12/02113
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Non-Small-Cell Lung Carcinoma; Digestive System Neoplasms; Breast Neoplasms
Keywords: physical exercise; Health Related Quality of Life; Non-Small-Cell Lung Carcinoma; digestive system neoplasms; breast neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Digestive System Neoplasms; Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise group (Experimental): supervised exercise program education program on healthy habits Pharmacological treatment and selfcare encouragement
  Interventions: Other: Supervised Physical activity; Behavioral: education program on healthy habits
- control group (No Intervention): Pharmacological treatment and selfcare encouragement.

INTERVENTIONS:
Other: Supervised Physical activity — Both groups received standardized usual care. The EP group will receive, in addition, a nurse supervised exercise program for 2 months in the PHC and a second phase in community facilities during the remaining 10 month
  Arms: Exercise group
Behavioral: education program on healthy habits — education program on healthy habits for 2 months in the PHC and a second phase in community facilities during the remaining 10 months
  Arms: Exercise group

SUMMARY:
AIM: To evaluate the effectiveness and efficiency of an innovative exercise program (EP) for patients during treatment for gastrointestinal tumors, breast and non small cells lung cancer, in terms of improved quality of life (QOL), fatigue and functional capacity respect the usual standard treatment (ST). DESIGN: Pragmatic randomized clinical trial in two parallel groups: EP and ST. SETTING: 7 Primary Health Centers (PHC) of the redIAPPISCIII, in coordination with oncology services. PARTICIPANTS: 250 patients with the above tumors, locally advanced or with metastatic disease, in adjuvant treatment, with Performance Status(PS) PS1-PS0. INTERVENTION: Both groups received standardized usual care. The EP group will receive, in addition, a nurse supervised exercise program for 2 months in the PHC and a second phase in community facilities during the remaining 10 months. MEASUREMENTS: The primary outcome measure is the change from baseline in the QOL+66 treatment, as measured by the specific questionnaire for patients with cancer EORTC QLQ-C-30 and Short Form(SF-36) overall. Secondary: fatigue (FACIT-F), radiological response, functional capacity (6 minutes walking and cardiopulmonary test), muscle strength and progression-free survival and overall. Predictors and confounders: age, sex, stage and tumor type, histology, treatment. ANALYSIS: We will compare between groups mean changes from baseline measurement of quality of life questionnaire (QOL) and other variables, on an intention to treat basis, using longitudinal mixed-effects models for repeated measures at 2, 6 and 12 months follow-up. Cost / effectiveness and cost / incremental utility associated to the program wil be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years
* Diagnosis of digestive system cancer , breast cancer or histologically confirmed NSCLC stage IV Physical Status (PS) 0 or 1.
* First-line chemotherapy treatment for each type of standard tumor
* Adequate renal, liver and blood function.

Exclusion Criteria:

* Brain metastases
* Risk of fracture (bone metastases)
* Unstable heart disease, uncontrolled BP Systolic Blood Pressure((SBP)> 200 or Diastolic Blood Pressure (DBP)> 110), heart failure (NYHA II or greater), constrictive pericarditis
* Other diseases at the discretion of the investigator to be a contraindication for physical exercise.
* Perform regular physical activity (150 minutes / week of moderate or vigorous 75)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-01 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Health Related Quality of Life (EORTC QLQ-C30) | basal,2,6,12 months fllow up

SECONDARY OUTCOMES:
asthenia measurement with FACIT-F (Functional Assessment of Chronic Illness Therapy-Fatigue) questionaire | Basal, 2,6 and12 months
Functional Capacity-6 minute Walking test | basal, 2,6 and 12 months
cardiorespiratory test | basal, 2, 6 and12 months
Changes in Muscular Strenght-Dynamometer | basal, 2,6 nad 12 months
progression-free survival | basal, 2, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: GRANDES GONZALO, Medicine, Principal Investigator — Primary Care Research Unit of Bizkaia (Basque Health Service); ARIETALEANIZBEASCOA MARIA SOLEDAD, NURSE, Study Director — Primary Care Research Unit of Bizkaia (Basque Health Service)
Locations (1):
- Primary Care Research Unit of Bizkaia, Bilbao, Bizkaia, Spain

REFERENCES:
- [Derived] Mendizabal-Gallastegui N, Arietaleanizbeaskoa MS, Latorre PM, Garcia-Alvarez A, Sancho A, Iruarrizaga E, Lopez-Vivanco G, Grandes G. Nurse-Supervised Exercise for People with Stage IV Cancer: The EFICANCER Randomized Clinical Trial. Semin Oncol Nurs. 2023 Aug;39(4):151448. doi: 10.1016/j.soncn.2023.151448. Epub 2023 May 13. PMID 37183104
- [Derived] Sancho A, Carrera S, Arietaleanizbeascoa M, Arce V, Gallastegui NM, Gine March A, Sanz-Guinea A, Eskisabel A, Rodriguez AL, Martin RA, Lopez-Vivanco G, Grandes G. Supervised physical exercise to improve the quality of life of cancer patients: the EFICANCER randomised controlled trial. BMC Cancer. 2015 Feb 6;15:40. doi: 10.1186/s12885-015-1055-x. PMID 25655792